CLINICAL TRIAL: NCT02965352
Title: Peripheral for Quantify Strength of Children Functional During the Pinch Movement
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Mogi das Cruzes (Other)
Responsible Party: Principal Investigator, Silvia Regina M. S. Boschi, PhD, University of Mogi das Cruzes
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 45883715.9.0000.5497
Record Dates: First submitted 2016-11-08; First posted 2016-11-16 (Estimated); Last update posted 2016-11-21 (Estimated); Status verified 2016-11

CONDITIONS: Hand Strength

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Hand strength (Experimental): Volunteers without motor abnormalities. The tests were performed in a single session lasting 30 minutes, when volunteers used the door handle device, the linear switch device, and the door key device, in order to quantify the hand strength.
  Interventions: Device: Door handle device; Device: Linear switch device; Device: Door key device

INTERVENTIONS:
Device: Door handle device — To evaluate the cylindrical grip movement, it was used a door handle, which evaluated all the strength at the arc of motion
Device: Linear switch device — To evaluate the pulp-pulp pinch movement, it was used one linear switch, which evaluated all the strength at the motion displacement.
Device: Door key device — To evaluate the pulp-side pinch movement, it was used a door key, which evaluated all the strength at the arc of motion

SUMMARY:
This study has developed a peripheral to quantify the functional strength of children without motor change during the movement of grip and pinch. It was possible to know the exact values of these strengths, the range of motion that was made, and also if the grip strength was maintained during all the arc of motion.

DETAILED DESCRIPTION:
Since childhood, it has been necessary to produce sufficient force to grip and pinch, for performing daily tasks independently; therefore, measurements of these forces end up being useful markers to evaluate the performance and the physical development of the child. It was developed a peripheral containing three devices and instrumented for analyzing the force applied during execution of the cylindrical grip movement, pinch pulp-side and pinch pulp-pulp in different situations of the daily life of the volunteer. The data acquisition interface was developed in a software for data recording. For the peripheral functionality tests, thirty volunteers of both genders were selected. They were also students of the Sports Secretary, with no motor abnormalities, between seven and ten years old.

ELIGIBILITY:
Inclusion Criteria:

* change Absence of skeletal muscle in the upper limbs
* neurological disorder Absence
* Informed Consent signed by the responsible
* with preserved cognitive.
* consent form signed by the volunteer

Exclusion Criteria:

* Having less than 7 years old
* Having more than 10 years old
* To present some compromise skeletal muscle in the upper limbs
* not take part in the research

Ages: 7 Years to 10 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2015-06; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
Force | 15 minutes
  The force of cylindrical grip movement was measured through a door handle device, pinch pulp-side through a door key and pinch pulp-pulp movement through a switch. The test was measured 3 times with 1 minute interval and it was measured the strength during all arc of motion. Unit of measurement: Newton (N).

SECONDARY OUTCOMES:
range of motion in angle | 15 minutes
  The test measured the range of motion in a door handle device and in a door key device 3 times with 1 minute interval for each test, in which all the range of motion was measured from its start until its end. Unit of measurement: Angle (º).
range of motion in percentage | 15 minutes
  The test measured the range of motion in a linear switch device 3 times with 1 minute interval for each test, in which all of the range of motion was measured from its start until its end. Unit measurement: Percentage (%).

CONTACTS AND LOCATIONS:
Overall Officials: Silvia R Boschi, PhD, Principal Investigator — University of Mogi das Cruzes

IPD SHARING:
Plan to Share IPD: Undecided